CLINICAL TRIAL: NCT03216252
Title: IMPLEMENTING A SINGLE MUSCLE FIBER DNA QUANTIFICATION TECHNIQUE AS A INTERPRETATION TOOL FOR THE VARIANTS OF UNKNOWN SERVICE IN MITOCHONDRIAL DISEASES
Brief Title: DNA QUANTIFICATION TECHNIQUE AS A INTERPRETATION TOOL IN MITOCHONDRIAL DISEASES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOIP-04
Record Dates: First submitted 2017-07-07; First posted 2017-07-13 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Mitochondrial Diseases
MeSH Terms: conditions — Mitochondrial Diseases | interventions — Sampling Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biological samples (Other): biological samples on patients with MITOCHONDRIAL DISEASES
  Interventions: Biological: samples

INTERVENTIONS:
Biological: samples — Blood samples, oral smear and urine

SUMMARY:
2622/5000 Mitochondrial diseases (MM) are the most common metabolic diseases. Since these pathologies are very heterogeneous in clinical terms, only the identification of mutations in nuclear genes or mitochondrial DNA confirms the diagnosis.

The full-scale study of mtDNA by high-throughput sequencing (NGS) is a first step in the diagnostic approach. The recent introduction of this revolutionary new technology has greatly increased the efficiency of mutation identification. However, in addition to known pathogenic mutations, NGS reveals numerous variants whose significance is currently unknown. A major challenge to obtain a reliable diagnosis is therefore the interpretation of the clinical impact of these new rare variants which proves to be very difficult.

Pathogenicity criteria allow the classification of variants from benign to pathogenic. One of the major pathogenicity criteria is a good correlation of heteroplasmic level with tissue or cellular involvement. Indeed, mtDNA mutations are generally heteroplasmic, which corresponds to the coexistence of normal and mutated molecules in the same cell or tissue, the most affected tissues having a high rate of mutation. On a muscle biopsy of an affected patient, the fibers often present an enzyme deficiency in cytochrome c oxidase (COX-negative) which can be demonstrated in immunohistochemistry. The single fiber study allows to isolate the deficient fibers and to quantify the heteroplasmic rate of a variant. The presence of a high level of heteroplasm in the COX-negative fibers, unlike fibers without deficit, is a strong argument in favor of the pathogenicity of this variant. Currently, this technique is not used routinely in diagnostic laboratories but only occasionally in a research framework in some laboratories. It is a heavy technique that consists of a first stage of laser microdissection of the various muscle fibers followed by a second step of quantification of the variant from each fiber. This second step requires a specific focus for each identified variant.

The aim of this pilot study is to develop a new technique for quantification of single-fiber heteroplasmics isolated by NGS laser microdissection. This, independent of the type of variant, will avoid the long and costly adjustments required for each new variant identified and thus facilitate its use

ELIGIBILITY:
Inclusion Criteria:

* general criteria: major or minor patients, sporadic or isolated cases
* criteria related to pathology:
* Suspected mitochondrial pathology which will be evaluated according to the following criteria (expertise of the clinician of the MM reference center):
* Clinical picture suggestive of a mitochondrial pathology ("illegitimate association" of symptoms, specific syndrome of MELAS type for example, muscular deficit, ptosis ...) AND / OR

  * Metabolic assessment suggestive of respiratory tract involvement AND / OR
  * Identification of a deficiency involving one or more complexes of the respiratory chain from a muscular specimen
* Presence on the histological analysis of the muscle biopsy of COX-negative fibers
* signing of informed consent for minor patients signed by at least one of the parents or the representative of the parental authority

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision;
* Persons hospitalized without consent;
* Persons admitted to a health or social institution for purposes other than research;
* Persons of legal age who are under protection or who are unable to express their consent. Inability to co-operate.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
number of amplification with the NGS technique | 36 months

SECONDARY OUTCOMES:
comparaison of the number of amplification between NGS technique and the PCR-RFLP technique | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No